CLINICAL TRIAL: NCT02114931
Title: An Open-label, Single-arm Extension Study to Evaluate the Long-term Safety and Efficacy of ABP 501 in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Long-term Safety and Efficacy of ABP 501 in Subjects With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20130258; 2013-004654-13 (EudraCT Number)
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: arthritis; rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — ABP 501; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABP 501 (Experimental): Participants received ABP 501 40 mg subcutaneously (SC) every other week for up to 18 months.
  Interventions: Biological: ABP 501

INTERVENTIONS:
Biological: ABP 501 — Solution for subcutaneous injection in a syringe containing 40 mg/0.8 mL ABP 501
  Other Names: AMJEVITA™; Adalimumab-atto

SUMMARY:
The purpose of this open-label study is to evaluate the long-term safety and efficacy of ABP 501 in adults with moderate to severe rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Subject was randomized into protocol 20120262 (NCT01970475) and completed the week 26 visit

Exclusion Criteria:

* Subject experienced a serious adverse event (SAE) or an adverse event (AE) in the 20120262 study that could cause extension treatment to be detrimental
* Subject completed study 20120262 but cannot be dosed within 4 weeks of the week 26 visit of study 20120262
* Current infection requiring the use of oral or intravenous antibiotics

Other Inclusion/Exclusion criteria may apply

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amgen MD, Study Director — Amgen
Locations (67):
- United States (29):
  - Research Site, Huntsville, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Covina, California
  - Research Site, El Cajon, California
  - Research Site, Hemet, California
  - Research Site, Palm Desert, California
  - Research Site, Van Nuys, California
  - Research Site, Whittier, California
  - Research Site, Danbury, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sandy Springs, Georgia
  - Research Site, Lexington, Kentucky
  - Research Site, Hagerstown, Maryland
  - Research Site, Wheaton, Maryland
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Brooklyn, New York
  - Research Site, Mineola, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, Spokane, Washington
- Bulgaria (3):
  - Research Site, Plovdiv, Plovdiv
  - Research Site, Rousse, Ruse
  - Research Site, Soifia, Sofia
- Canada (3):
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Windsor, Ontario
- Czechia (5):
  - Research Site, Prague, Prague
  - Research Site, Hlučín, Severomoravsky Kraj
  - Research Site, Ostrava, Severomoravsky Kraj
  - Research Site, Zlín, Severomoravsky Kraj
  - Research Site, Prague
- Germany (4):
  - Research Site, Hamburg, Hamburg
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Ratingen, North Rhine-Westphalia
  - Research Site, Leipzig, Saxony
- Hungary (4):
  - Research Site, Budapest, Budapest
  - Research Site, Szentes, Csongrád megye
  - Research Site, Balatonfüred, Veszprém megye
  - Research Site, Veszprém, Veszprém megye
- Poland (12):
  - Research Site, Kościan, Greater Poland Voivodeship
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Torun, Kuyavian-Pomeranian Voivodeship
  - Research Site, Wroclaw, Lower Silesian Voivodeship
  - Research Site, Lublin, Lublin Voivodeship
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Gdynia, Pomeranian Voivodeship
  - Research Site, Działdowo, Warmian-Masurian Voivodeship
  - Research Site, Elblag, Warmian-Masurian Voivodeship
- Research Site, Brăila, Brăila County, Romania
- Research Site, Petrozavodsk, Russia
- Spain (4):
  - Research Site, Santiago de Compostela, A Coruna
  - Research Site, A Coruña, La Coruna
  - Research Site, Madrid, Madrid
  - Research Site, Seville, Sevilla
- Research Site, Suffolk, England, United Kingdom

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165
- [Derived] Cohen S, Pablos JL, Pavelka K, Muller GA, Matsumoto A, Kivitz A, Wang H, Krishnan E. An open-label extension study to demonstrate long-term safety and efficacy of ABP 501 in patients with rheumatoid arthritis. Arthritis Res Ther. 2019 Mar 29;21(1):84. doi: 10.1186/s13075-019-1857-3. PMID 30922373
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 83 centers in 11 countries in Eastern Europe, North America and Western Europe.
Pre-assignment Details: Study 20130258 was a single-arm, open-label extension of the parent Study 20120262 (NCT01970475). Results are reported according to treatment in the parent Study 20120262.
Groups:
- ABP 501/ABP 501: Participants who received ABP 501 in the parent study continued to receive ABP 501 40 mg subcutaneously (SC) every other week for an additional 18 months (total of 24-months treatment).
- Adalimumab/ABP 501: Participants who received adalimumab in the parent study transitioned to receive ABP 501 40 mg subcutaneously every other week for 18 months.
Period: Overall Study
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Started | 230 | 237
Received Treatment | 229 (One participant was enrolled in error and did not receive treatment in the extension study) | 237
Completed | 205 | 207
Not Completed | 25 | 30
Not completed — Withdrawal by Subject | 15 | 18
Not completed — Adverse Event | 4 | 6
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 1 | 2
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501 | Total
Number analyzed (Participants) | 230 | 237 | 467
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at baseline of parent study
  years | 54.7 (11.71) | 56.1 (11.40) | 55.4 (11.56)
Age, Customized [Number; unit: participants] — Age at baseline of parent study
  participants
    Between 18 and 65 years | 183 | 181 | 364
    ≥ 65 years | 47 | 56 | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 188 | 191 | 379
  Male | 42 | 46 | 88
Race/Ethnicity, Customized [Number; unit: participants]
  White | 218 | 224 | 442
  Black or African American | 8 | 12 | 20
  Asian | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Mixed Race | 0 | 0 | 0
  Other | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 27 | 19 | 46
  Not Hispanic or Latino | 202 | 217 | 419
  Not Allowed to Collect | 1 | 1 | 2
Geographic Region [Number; unit: participants]
  Eastern Europe | 153 | 156 | 309
  Western Europe | 12 | 19 | 31
  North America | 65 | 62 | 127
  Latin America | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 according to the following scale:
  1 = mild; 2 = moderate; 3 = severe; 4 = life-threatening; 5 = fatal. A treatment-related AE is defined as an event where the answer to the question "is there a reasonable possibility that the event may have been caused by the Investigational Medicinal Product" was yes.
  A serious adverse event is defined as an AE that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening (places the subject at immediate risk of death)
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event.
Time Frame: From the first dose of study drug in the extension study to 28 days following the last dose; 72 weeks
Population: The safety analysis set included all participants enrolled and treated with at least 1 dose of ABP 501 in the extension study.
Measure: Number; unit: participants
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Number analyzed (Participants) | 229 | 237
participants
  Any adverse event (AE) | 143 | 154
  Any grade ≥ 3 adverse event | 26 | 16
  Any treatment-related adverse event (TRAE) | 37 | 43
  Any grade ≥ 3 treatment-related adverse event | 3 | 4
  Any adverse event with outcome of death | 0 | 0
  Any TRAE with an outcome of death | 0 | 0
  Any serious adverse event (SAE) | 25 | 21
  Any treatment-related serious adverse event | 2 | 1
  Any AE leading to discontinuation of ABP 501 | 7 | 10
  Any TRAE leading to discontinuation of ABP 501 | 4 | 5
  Any AE leading to discontinuation from study | 3 | 5
  Any TRAE leading to discontinuation from study | 1 | 3

2. Primary Outcome: Number of Participants With Grade ≥ 3 Hematology and Chemistry Laboratory Results
Description: Laboratory results were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 according to the following scale:
  1 = mild; 2 = moderate; 3 = severe; 4 = life-threatening; 5 = fatal.
Time Frame: From the first dose of study drug in the extension study to 28 days following the last dose; 72 weeks
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Number analyzed (Participants) | 229 | 237
participants
  Hemoglobin (anemia) | 1 | 0
  Alanine aminotransferase (ALT) | 1 | 0
  Aspartate aminotransferase (AST) | 1 | 0
  Bilirubin | 1 | 0
  Gamma glutamyl transferase | 7 | 3
  Potassium (hyperkalemia) | 1 | 1

3. Primary Outcome: Percentage of Participants Who Developed Antibodies to ABP 501
Description: Two validated assays were used to detect the presence of anti-drug antibodies. All samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect anti-drug antibodies against ABP 501 (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a non-cell based bioassay to determine neutralizing activity against ABP 501. If a sample was positive for binding antibodies and demonstrated neutralizing activity at the same time point, the sample was defined as positive for neutralizing antibodies.
  Preexisting antibody positive indicates participants with a positive result at baseline of the extension study. Developing antibody positive indicates participants with a negative or no result at baseline of the extension study who were positive at any time point post-baseline during the extension study.
Time Frame: Up to week 72
Population: The anti-drug antibody analysis set includes participants who received at least 1 dose of ABP 501 in the extension study and who had at least 1 evaluable antibody test assay against ABP 501 in the extension study.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Number analyzed (Participants) | 229 | 237
percentage of participants
  Preexisting Binding Antibody Positive | 32.3 | 34.2
  Preexisting Neutralizing Antibody Positive | 5.7 | 8.9
  Developing Binding Antibody Positive | 21.8 | 14.8
  Developing Neutralizing Antibody Positive | 8.7 | 5.1

4. Secondary Outcome: Percentage of Participants With an American College of Rheumatology (ACR) 20 Response
Description: A participant was a responder if the following 3 criteria for improvement from Baseline of the parent study were met:
  * ≥ 20% improvement in tender joint count;
  * ≥ 20% improvement in swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-Reactive Protein level.
Time Frame: Parent study baseline, extension study baseline and weeks 4, 24, 48, and 70
Population: The full analysis set (all participants enrolled in the extension study) with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Number analyzed (Participants) | 230 | 237
percentage of participants
  Extension study baseline (n = 228, 236) | 73.2 | 73.3
  Week 4 (n = 228, 237) | 77.6 | 77.6
  Week 24 (n = 223, 230) | 74.0 | 74.3
  Week 48 (n = 216, 218) | 76.9 | 78.4
  Week 70 (n = 206, 209) | 79.6 | 78.0

5. Secondary Outcome: Change From Parent Study Baseline in Disease Activity Score 28-C-reactive Protein (DAS28-CRP)
Description: The DAS28-CRP is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP) level
  * Patient's global assessment of disease activity assessed on a score from 0 to 100 transformed from the result measured on a horizontal scale from 0 (no RA activity at all) to 10 (worst RA activity imaginable).
  The DAS28-CRP score ranges from approximately zero to ten. Higher DAS28-CRP scores indicate higher disease activity.
Time Frame: Parent study baseline, extension study baseline and weeks 4, 24, 48 and 70
Population: Full analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Number analyzed (Participants) | 230 | 237
units on a scale
  Extension Study Baseline (n = 219, 221) | -2.26 (1.255) | -2.25 (1.289)
  Week 4 (n = 228, 235) | -2.40 (1.322) | -2.32 (1.257)
  Week 24 (n = 223, 227) | -2.49 (1.272) | -2.33 (1.316)
  Week 48 (n = 216, 217) | -2.59 (1.433) | -2.51 (1.414)
  Week 70 (n = 205, 207) | -2.70 (1.389) | -2.51 (1.445)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug in the extension study to 28 days following the last dose; 72 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | ABP 501/ABP 501 | Adalimumab/ABP 501
Serious Adverse Events (participants affected / at risk) | 25/229 | 21/237
Other Adverse Events (participants affected / at risk) | 72/229 | 71/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 501/ABP 501 (N=229) | Adalimumab/ABP 501 (N=237)
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 2
Macular degeneration (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Device failure (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Uterine cervical erosion (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bunion operation (Surgical and medical procedures) | 0 | 1
Prosthesis implantation (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABP 501/ABP 501 (N=229) | Adalimumab/ABP 501 (N=237)
Bronchitis (Infections and infestations) | 16 | 13
Nasopharyngitis (Infections and infestations) | 18 | 25
Pharyngitis (Infections and infestations) | 12 | 7
Upper respiratory tract infection (Infections and infestations) | 18 | 22
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11 | 17
Hypertension (Vascular disorders) | 16 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.